CLINICAL TRIAL: NCT02633098
Title: Phase II Randomised, Double Blind, Placebo Controlled Trial of Neoadjuvant Artesunate in Stage II/III Colorectal Cancer
Brief Title: A Safety and Effectiveness Study of Pre-operative Artesunate in Stage II/III Colorectal Cancer
Acronym: NeoART
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: St George's, University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15.0154
Record Dates: First submitted 2015-11-18; First posted 2015-12-17 (Estimated); Last update posted 2022-10-12 (Actual); Status verified 2021-10

CONDITIONS: Colorectal Cancer; Bowel Cancer
Keywords: Artesunate; Artemisinins; Antimalarial; Neoadjuvant; Pre-operative
MeSH Terms: conditions — Colorectal Neoplasms; Intestinal Neoplasms | interventions — Artesunate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Artesunate (Experimental): Artesunate 200mg oral tablets once daily for 14 days.
  Interventions: Drug: Artesunate 200mg
- Matching placebo (Placebo Comparator): Matching placebo oral tablets once daily for 14 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Artesunate 200mg — Artesunate 200mg PO OD for 14 days prior to colorectal resection surgery
  Arms: Artesunate
Drug: Placebo — Matched placebo PO OD for 14 days prior to colorectal resection surgery
  Arms: Matching placebo

SUMMARY:
This study evaluates the safety and effectiveness of pre-operative artesunate given orally once a day for 14 days prior to surgery in patients with Stage II/III colorectal cancer.

Artesunate is an established antimalarial drug with an excellent safety profile, is well tolerated and affordable. A number of laboratory studies and one small pilot clinical study in patients with colorectal cancer have shown that artesunate can reduce the proliferation and growth of cancer cells.

Two hundred patients diagnosed with Stage II/III operable colorectal cancer will be randomly allocated to receive oral artesunate 200mg daily or a matching placebo for 14 days prior to surgery. Patients will be followed up closely for 5 years to see if giving artesunate preoperatively reduces the risk of cancer recurring after surgery.

DETAILED DESCRIPTION:
Artesunate is an established antimalarial drug belonging to the artemisinin class of drugs, has an excellent safety profile, is well tolerated and affordable. In last two decades, artemisinins have shown potent and broad anticancer properties in a range of cell lines and animal models, supporting the hypothesis that artemisinins have the potential to be an effective anti-cancer therapy. Multiple potential mechanisms of action include anti-proliferative effects through cell-cycle disruption, reactive oxygen species (ROS) -induced DNA damage, induction of apoptosis, anti-angiogenesis, immunomodulation and induced radiosensitivity.

Despite a multi-modality treatment approach to colorectal cancer, 5 year overall survival does not currently exceed 60%. Neoadjuvant pre-operative therapy may be more effective at eradicating micrometastases compared to adjuvant therapy delivered following the delay and immunological stress of surgery. However current neoadjuvant chemotherapy regimens are often associated with significant side effects and may result in a delay in surgery whilst patients recover. A well tolerated, affordable, novel anticancer agent that could be given to patients whilst they wait for surgery, without causing a surgical delay due to treatment related toxicity, would have a significant clinical impact on patient care.

The NeoART trial is a phase II multicentre randomised, double blind, placebo controlled trial (RCT) for patients undergoing primary surgery for Stage II/III colorectal cancers. Patients are randomised (1:1 ratio) to receive either a two week course of neoadjuvant artesunate 200mg once daily or matching placebo. Both patients and health care professionals are blinded to treatment allocation arm to minimise outcome-reporting bias. The primary endpoint of the trial is recurrence free survival two years after surgery. Secondary endpoints include 2 and 5 year overall survival, treatment related toxicity, tolerability and patient quality of life. A translational sub-study looking at predictive and prognostic biomarkers is also planned.

ELIGIBILITY:
Inclusion criteria

1. Aged 18 or over
2. Histologically proven single primary site colorectal adenocarcinoma or high grade dysplasia plus unequivocal radiological evidence of invasive cancer
3. Stage II/III colorectal cancer planned for surgical resection and no clinical indication for neoadjuvant preoperative chemotherapy/chemoradiation therapy
4. WHO performance status 0,1 or 2
5. Adequate full blood count: White Cell Count (WCC) >3.0 x 10^9 /l; Platelets >100 x 10^9/l; Haemoglobin (Hb) >80g/L
6. Adequate renal function: Glomerular Filtration Rate >30ml/min by Cockcroft-Gault formula
7. Adequate hepatobiliary function : Bilirubin < 3 x Upper limit normal
8. Female participants of child bearing potential must have a negative pregnancy test < 72 hours prior to initiating study intervention and agree to avoid pregnancy using adequate, medically approved contraceptive precautions for up to 6 weeks after the last dose of study treatment intervention
9. Male participants with a partner of childbearing potential must agree to use adequate, medically approved contraceptive precautions during and for up to 6 weeks after the last dose of the study treatment intervention
10. Patient able and willing to provide written, informed consent for the study.

Exclusion criteria

1. Contraindication to the use of artesunate due to hypersensitivity
2. Pregnancy or lactation
3. Male or female participants unwilling to use an effective method of birth control (either hormonal in the form of contraceptive pill or barrier method of birth control accompanied by the use of a proprietary spermicidal foam/gel or film); or agreement of true abstinence from time to consent is signed until 6 weeks after the last dose of study treatment intervention (i.e. withdrawal, calendar, ovulation, symptothermal and post ovulation methods are not considered acceptable methods)
4. History of immunosuppression
5. History of hearing or balance problems
6. Weight < 52kg or > 110kg
7. Other planned intervention, apart from standard of care
8. Any other malignant disease diagnosis within the preceding 2 years with the exception of non-melanomatous skin cancer and carcinoma in situ
9. Lactose intolerance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-04-26 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence free survival at 2 years | 2 years following study randomisation.

SECONDARY OUTCOMES:
Recurrence free survival at 5 years | 5 years from study randomisation
Overall survival at 2 and 5 years | 2 and 5 years from study randomisation
Colon cancer specific death at 2 and 5 years | 2 and 5 years from study randomisation
Number of patients experiencing artesunate drug related toxicity as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v4.0 | Assessment at Day 7 following start of study intervention (artesunate/matching placebo)
Number of patients experiencing artesunate drug related toxicity as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v4.0 | Assessment at Day 14 following start of study intervention (artesunate/matching placebo)
Number of patients experiencing artesunate drug related toxicity as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v4.0 | Assessment at Day 42 following start of study intervention (artesunate/matching placebo)
Adverse events affecting patients as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v4.0 | Assessment at Day 7 following study intervention
Adverse events affecting patients as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v4.0 | Assessment at Day 14 following study intervention
Adverse events affecting patients as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v4.0 | Assessment at Day 42 following study intervention
Adverse events affecting patients as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v4.0 | Assessment 6 months following study intervention
Adverse events affecting patients as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v4.0 | Assessment 12 months following study intervention
Adverse events affecting patients as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v4.0 | Assessment 18 months following study intervention
Adverse events affecting patients as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v4.0 | Assessment 24 months following study intervention
Adverse events affecting patients as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v4.0 | Assessment 30 months following study intervention
Adverse events affecting patients as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v4.0 | Assessment 36 months following study intervention
Adverse events affecting patients as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v4.0 | Assessment 42 months following study intervention
Adverse events affecting patients as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v4.0 | Assessment 48 months following study intervention
Adverse events affecting patients as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v4.0 | Assessment 54 months following study intervention
Adverse events affecting patients as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v4.0 | Assessment 60 months following study intervention
Pathological assessment of tumour regression (involvement of lymph nodes; serosa; resection margin) | Post surgical pathology review (following Day 14 of study intervention)
Patient quality of life | Assessment at Day 1 of study intervention
  Using validated quality of life self-administered questionnaires
Patient quality of life | Assessment at Day 7 of study intervention
  Using validated quality of life self-administered questionnaires
Patient quality of life | Assessment at Day 14 of study intervention
  Using validated quality of life self-administered questionnaires
Patient quality of life | Assessment at Day 42 of study intervention
  Using validated quality of life self-administered questionnaires
Surgical complications | From time of surgery up to 3 months post surgery
  Number of patients with surgery related adverse events as assessed by CTCAE v4.0
Predictive value of tumour marker Carcinoma Embryonic Antigen (CEA) kinetics in terms of predicting response to artesunate therapy | Assessment at Day 1 of study intervention
Predictive value of tumour marker Carcinoma Embryonic Antigen (CEA) kinetics in terms of predicting response to artesunate therapy | Assessment at Day 7 of study intervention
Predictive value of tumour marker Carcinoma Embryonic Antigen (CEA) kinetics in terms of predicting response to artesunate therapy | Assessment at Day 14 of study intervention
Predictive value of tumour marker Carcinoma Embryonic Antigen (CEA) kinetics in terms of predicting response to artesunate therapy | Assessment at Day 42 of study intervention
Immunohistochemical analyses of paraffin-embedded tumour sections to assess Kirsten rat sarcoma viral oncogene homolog (Kras) mutation status | Pre and post intervention tumour samples from patients (Day 0 and Day 15)
  Number of patients with Kras mutant tumours
Immunohistochemical analyses of paraffin-embedded tumour sections to assess Mismatch Repair (MMR) status | Pre and post intervention tumour samples from patients (Day 0 and Day 15)
  Number of patients with Mismatch Repair (MMR) mutant tumours
Immunohistochemical analyses of paraffin-embedded tumour for v-Raf murine sarcoma viral oncogene homolog B (BRAF) mutation status | Pre and post intervention tumour samples from patients (Day 0 and Day 15)
  Number of patients with BRAF mutant tumours
Immunohistochemical analyses of paraffin-embedded tumour for Platelet derived growth factor (PDGF) expression | Pre and post intervention tumour samples from patients (Day 0 and Day 15)
  Number of patients whose tumours show PDGF upregulation/downregulation following treatment intervention
Immunohistochemical analyses of paraffin-embedded tumour for Platelet derived growth factor receptor (PDGFR) expression | Pre and post intervention tumour samples from patients (Day 0 and Day 15)
  Number of patients whose tumours show PDGFR upregulation/downregulation following study intervention
Immunohistochemical analyses of paraffin-embedded tumour for Vascular endothelial Growth Factor (VEGF) expression | Pre and post intervention tumour samples from patients (Day 0 and Day 15)
  Number of patients whose tumours show VEGF upregulation/downregulation following study intervention
Immunohistochemical analyses of paraffin-embedded tumour on Vascular endothelial Growth Factor Receptor (VEGFR) expression | Pre and post intervention tumour samples from patients (Day 0 and Day 15)
  Number of patients whose tumours show VEGFR upregulation/downregulation following study intervention
Determination of proliferative activity (Ki-67 staining, Cluster of Differentiation 31 protein (CD31) staining) | Pre and post intervention tumour samples from patients (Day 0 and Day 15)
  Number of patients whose tumours show an increase or reduction in proliferation markers Ki67 and CD31 following study intervention
Determination of activation of the Deoxyribonucleic acid damage response (DDR) pathway | Pre and post intervention tumour samples from patients (Day 0 and Day 15)
  Number of patients whose tumour samples show activation of the DDR pathway following study intervention
Wnt/β-catenin proliferation pathway protein expression (e.g. c-myc and cyclinD1 proteins) | Pre and post intervention tumour samples from patients (Day 0 and Day 15)
  Number of patients who show an increase or a decrease in expression of proteins involved in the Wnt/β-catenin proliferation pathway (e.g. c-myc and cyclinD1 proteins) following study intervention

CONTACTS AND LOCATIONS:
Overall Officials: Professor Sanjeev Krishna, BMBCh, DPhil, ScD, Principal Investigator — St George's University Hospitals NHS Foundation Trust
Locations (8):
- United Kingdom (8):
  - Medway Maritime Hospital, Gillingham, Kent
  - Kent Oncology Centre, Maidstone Hospital, Maidstone, Kent
  - Barking, Havering and Redbridge University Hospitals NHS Trust, Barking
  - Ashford & St Peters Hospital NHS Foundation Trust, Chertsey
  - University Hospitals of Derby and Burton NHS Foundation Trust, Derby
  - St George's University Hospitals NHS Fundation Trust, London
  - Norfolk & Norwich University Hospitlas NHS FT, Norwich
  - Shrewsbury and Telford Hospital NHS Trust, Shrewsbury